CLINICAL TRIAL: NCT02259166
Title: Impact of the Evaluation of the Enhanced Homestead Food Production Program in Sengerema, and Ukerewe in the Lake Zone,Tanzania
Brief Title: Enhanced Homestead Food Production Plus+ Program in the Lake Zone, Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Helen Keller International (Other); Foreign Affairs, Trade and Development, Canada (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EHFP+ TZ
Record Dates: First submitted 2014-09-05; First posted 2014-10-08 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2015-09

CONDITIONS: Anemia; Growth Retardation
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EHFP+ (Experimental): Group receiving the intervention EHFP+, in addition to MNPs distribution for 2 months and malaria diagnosis and treatment for children enrolled, at baseline and after 12 months
  Interventions: Other: EHFP+
- Control (No Intervention): MNPs distribution for 2 months and malaria diagnosis and treatment for children enrolled, at baseline and after 12 months

INTERVENTIONS:
Other: EHFP+ — Enhanced-homestead food production program including home gardening and poultry rearing + WASH interventions + SBCC around the essential nutrition actions and WASH/malaria prevention with a gender component.
  Arms: EHFP+

SUMMARY:
The purpose of this study is to assess if the Enhanced Homestead Food Production Plus (EHFP+) Program implemented by HKI in Mwanza, Tanzania, enhances uptake of Micronutrient Powder (MNP) supplementation in children, helps maintaining reduced anemia levels among children after a blanket provision of MNP, and has an impact on child growth, infant and young child feeding (IYCF) practices, maternal knowledge related to health, nutrition, WASH and malaria prevention, food security and women's empowerment.

DETAILED DESCRIPTION:
Since 1988, Helen Keller International's (HKI) flagship Homestead Food Production (HFP) program in Asia has helped communities establish technically-improved local food production systems by creating gardens yielding micronutrient-rich fruits and vegetables over expanded growing seasons, complemented by the improved rearing of poultry and livestock.

In 2010, HKI introduced an enhanced-HFP (E-HFP) model in Burkina Faso and included a strengthened nutrition education component; the Essential Nutrition Actions (ENA) framework. This E-HFP program was evaluated by IFPRI and yielded some encouraging results. With regards to nutritional outcomes, however, the primary finding was that, while the E-HFP program improved hemoglobin concentration-an indicator of iron status-the evaluation failed to note a significant impact of the program on improving children's growth. The primary explanation for the absence of a measurable improvement in children's growth was the lack of complementary health interventions that aim to specifically reduce children's disease burden, which, along with the lack of adequate food and care, is an underlying cause of undernutriton (UNICEF 1990).

Building on lessons learned from the Burkina Faso E-HFP program and a 2011 Tanzania HFP program, a new model, the Enhanced Homestead Food Production Plus (E-HFP+), was developed for Tanzania to improve the nutritional status of infants and young children. The new model strengthens the Behavior Change Communication (BCC) on malaria prevention, WASH, and gender components and enhances links with the health sector. The model will also test two new concepts:

1. to assess if the E-HFP+ program has the potential to maintain adequate levels of hemoglobin concentrations by increasing iron-rich food consumption and malaria prevention good practices.
2. to assess the effectiveness on anemia of using an existing agriculture-based platform to promote uptake and utilization of MNP.

The model involves both a set of production and nutrition interventions targeted to mothers and the provision of a curative treatment for moderate to severe anemia (Micronutrient Powder).

The main objective of the impact evaluation of the E-HFP+ program is therefore to assess whether the program:

* Maintains reduced anemia levels among pre-school aged children after a blanket provision of Micronutrient Powder (MNP)
* Improves child growth (measured by HAZ and WHZ)
* Improves infant and young child feeding (IYCF) practices and maternal knowledge on health and nutrition
* Is an appropriate delivery platform to enhance uptake and utilization of MNP supplementation in children

ELIGIBILITY:
Inclusion Criteria:

* women living in the study area
* having one child aged 6-12 months of age

Exclusion Criteria:

* children with severe anemia

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2325 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Anemia (g/dl and %) | Measurements will be made for children aged 6 to 11 months at baseline and up to 3 months, 6 months, 12 months and 18 months (at endline), when the children are between the ages of 24 and 30 months
  Change in prevalence of anemia and hemoglobin concentration will be measured over the course of the program period.(at baseline, during follow-up after 3, 6 and 12 months and after 18 months at endline)

SECONDARY OUTCOMES:
Growth (Z-score and %) | Measurements will be made for children between the ages of 6 and 11 months of age at baseline and 18 months later, at endline, when the children are between the ages of 24 and 30 months
  Change in height-for-age Z-scores, weight-for-age Z-scores and weight-for-height Z-scores will be measured as well as the change in the prevalence of stunting (HAZ<-2), underweight (WAZ<-2) and wasting (WHZ<-2) over the course of the program period
Biochemical markers | Baseline (June 2014), Follow-up1 (up to 3 months) and after 18 months at Endline
  Change in plasmatic concentration of iron biomarkers (transferring receptors and ferritin; TfR and F), in concentration of vitamin A biomarkers (retinolbindingprotein; RBP) and inflammatory proteins (C-reactiveprotein and alpha-1 acidglycoprotein; CRP and AGP)
Dietary diversity (%) | Baseline (2014) and after 18 months at Endline
  Measured with a questionnaire using a qualitative 24h recall. Unit: Number of food group consumed and percentage of children having consumed 4 groups (upon 7) the previous day
Food security (%) | Baseline (2014) and after 18 months at Endline (2016)
  Measured with a questionnaire to calculate the HFIAS score. Unit: percentage of household
Women's empowerment (%) | Baseline (2014) and after 18 months at Endline (2016)
  Measured by questionnaire, using a decision-making module and a domestic violence module. Percentage of women over a calculated score.
Maternal health and nutrition/WASH/malaria-related knowledge (%) | Baseline (2014) and after 18 months at Endline (2016)
  Using questionnaire on knowledge. Percentage of women giving adequate answer.
IYCF/WASH/malaria practices (%) | Baseline (2014) and after 18 months at Endline (2016)
  Using questionnaire on practices. Percentage of women with adequate practices.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Rawat, PhD, Principal Investigator — International Food Policy Research Institute; Erin Smith, Principal Investigator — Helen Keller International
Locations (1):
- National Institute for Medical Research, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: No